CLINICAL TRIAL: NCT04581187
Title: An onLine-pLatform to Improve Patient-centered Care During the COVID-19 pAndemic: a GIMEMA surveillaNce Program in hematologiC malignanciEs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: GIMEMA-ALLIANCE Platform
Record Dates: First submitted 2020-09-30; First posted 2020-10-09 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life assessment — Quality of life questionnaires

SUMMARY:
This is a national multicenter prospective observational study led by the GIMEMA. The GIMEMA-ALLIANCE Platform is also an online monitoring system for patients with hematologic malignancies aiming at helping hematologists in the early recognition and timely management of problems of their patients. Based on patient's rating of specific items (i.e. on the presence of clinically relevant problems or problems with adherence to therapy or risk of SARS-CoV-2 infection), the Platform will automatically send alerts to the treating hematologist (and/or appointed members of the local Team). Physicians will be free to make any action they feel appropriate for the best care of their patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any hematologic malignancy according to 2016 WHO classification
* Adult Patients (≥18 years).
* Written informed consent

Exclusion Criteria:

* Major cognitive deficits or psychiatric problems hampering a self-reported evaluation.
* Not able to read and understand local language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with any hematologic malignancy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HRQOL in adult patients with hematologic malignancies | After 2 years from date of registration
  To prospectively assess HRQOL in adult patients with hematologic malignancies, overall and by patient subgroups (e.g., by diagnosis of COVID-19)
Symptoms in adult patients with hematologic malignancies | After 2 years from date of registration
  To prospectively assess symptoms in adult patients with hematologic malignancies, overall and by patient subgroups (e.g., by diagnosis of COVID-19)
Adherence to therapy in adult patients with hematologic malignancies | After 2 years from date of registration
  To prospectively assess adherence to therapy in adult patients with hematologic malignancies, overall and by patient subgroups (e.g., by diagnosis of COVID-19)

SECONDARY OUTCOMES:
Prevalence of clinically relevant functional limitations and symptoms | After 2 years from date of registration
  To describe the prevalence of clinically relevant functional limitations (e.g., physical and social) and symptoms (e.g., fatigue, pain and dyspnea) by type of hematologic malignancy and by type of treatment (e.g., standard chemotherapy of oral anticancer therapies)
Factors associated with physical and mental health concerns, as measured by EORTC QLQ-C30 questionnaire | After 2 years from date of registration
  To investigate factors associated with physical and mental health concerns
Financial and social impact imposed by the COVID-19 pandemic on patient health outcomes | After 2 years from date of registration
  To examine the financial and social impact imposed by the COVID-19 pandemic on patient health outcomes
Limitations in accessing routine medical care services imposed by the COVID-19 pandemic on patient health outcomes | After 2 years from date of registration
  To examine the limitations in accessing routine medical care services imposed by the COVID-19 pandemic on patient health outcomes
Clinical strategies adopted by physicians | After 2 years from date of registration
  To describe clinical strategies adopted by physicians in response to patient-generated alerts, across different clinical scenarios

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vignetti, Principal Investigator — GIMEMA Foundation
Locations (27):
- Italy (27):
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona, Ancona
  - Irccs Centro Di Riferimento Oncologico Di Aviano - Sosd Oncoematologia Trapianti Emopoietici E Terapie Cellulari, Aviano
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Irccs Oncologico Istituto Tumori Giovanni Paolo II - UO Ematologia, Bari
  - Asl Della Provincia Di Barletta, Andria, Trani, Ospedale "Mons. Dimiccoli" - UOC Ematologia, Barletta
  - AO Brotzu, Presidio Ospedaliero A. Businco - Cagliari - SC Ematologia E CTMO, Cagliari
  - Aou Policlinico Vittorio Emanuele, Presidio Ospedaliero Ferrarotto -Divisione Clinicizzata Di Ematologia, Catania
  - Aou Ospedali Riuniti - Foggia- UOC Ematologia, Foggia
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Aou Di Modena- Sc Ematologia- Dipartimento Di Oncologia Ed Ematologia, Modena
  - Ao Di Rilievo Nazionale Antonio Cardarelli - UOC Ematologia, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Aou Maggiore Della Carità Di Novara, Novara
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Aou Policlinico P. Giaccone - Uo Ematologia Dipartimento Biomedico Di Medicina Interna E Specialistica, Palermo
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Ausl Reggio Emilia, Presidio Ospedaliero "Arcispedale Santa Maria Nuova" - Irccs- Uo Ematologia, Reggio Emilia
  - Ao San Camillo Forlanini - Uoc Ematologia E Trapianto Cellule Staminali, Roma
  - AOU Policlinico Tor Vergata - UOC Trapianto Cellule Staminali, Roma
  - Aou Policlinico Umberto I - Dipartimento Di Medicina Traslazionale - Sezione Ematologia, Roma
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Divisione di Ematologia - Ospedale S. Eugenio, Roma
  - Policlinico Universitario Campus Bio Medico - Roma - Uoc Ematologia E Trapianto Di Cellule Staminali, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari
  - Ospedale Di Sassuolo Spa - Ematologia, Sassuolo
  - Asl To 2, Torino Nord Emergenza San Giovanni Bosco - Ssd Ematologia, Torino
  - Torino Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino

REFERENCES:
- [Derived] Efficace F, Breccia M, Fazi P, Cottone F, Holzner B, Vignetti M. The GIMEMA-ALLIANCE Digital Health Platform for Patients With Hematologic Malignancies in the COVID-19 Pandemic and Postpandemic Era: Protocol for a Multicenter, Prospective, Observational Study. JMIR Res Protoc. 2021 Jun 1;10(6):e25271. doi: 10.2196/25271. PMID 33890580